CLINICAL TRIAL: NCT05808322
Title: An Open Label, Control Study to Evaluate the Efficacy and Safety of Ropeginterferon Alfa-2b in Adult COVID-19 Patients With Comorbidities
Brief Title: Clinical Study for the Efficacy and Safety of Ropeginterferon Alfa-2b in Adult COVID-19 Patients With Comorbidities
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202302136MIP-1
Record Dates: First submitted 2023-04-09; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Treated with P1101 (Ropeginterferon alfa-2b) plus standard of care (SOC)
  Interventions: Drug: Ropeginterferon alfa-2b; Procedure: SOC
- Control Group (Active Comparator): Treated with SOC alone
  Interventions: Procedure: SOC

INTERVENTIONS:
Drug: Ropeginterferon alfa-2b — A maximum of 3 doses of ropeginterferon alfa-2b will be given biweekly during the whole study period. A single dose of 250 μg ropeginterferon alfa-2b will be subcutaneous administrated at Day 1 visit. SARS-CoV-2 antigen test will be conducted at D15 and D29 visits. For patients who still have positive result in SARS-CoV-2 antigen test at Day 15 visit, the second dose of ropeginterferon alfa-2b at 350 μg will be subsequently administered at Day 15 visit. For patients who still have positive result in SARS-CoV-2 antigen test at Day 29 visit, the third dose of ropeginterferon alfa-2b at 500 μg will be administered at Day 29 visit.
  Other Names: P1101
  Arms: Study Group
Procedure: SOC — SOC includes infection prevention and control measures, supportive care, dexamethasone, and antiviral agents. The SOC is based on the Taiwan Centers for Disease Control (CDC) guidance and investigator's discretion.

SUMMARY:
To evaluate the efficacy of subcutaneous ropeginterferon alfa 2b ( P1101 combined with standard of care (SOC) compared with standard care alone in adult COVID-19 patients with comorbidities.

DETAILED DESCRIPTION:
This is a multi-center, open label, control study to evaluate the efficacy and safety of ropeginterferon alfa-2b in the treatment of adult COVID-19 patients with comorbidities. Adult COVID-19 patient with the specific comorbidities and being non-responder to the other anti-SARS-CoV-2 drugs, i.e., remdesivir, nirmatrelvir/ritonavir, and molnupiravir, or the patients who is not suitable to receive the other anti-SARS-CoV-2 drugs by investigator's judgement and has positive result (Ct <30) 14 days after the symptom onset of COVID-19 will be enrolled. The eligible patients will be randomized to receive the ropeginterferon alfa-2b plus SOC (study group) or to receive SOC alone (control group). For study group, a single dose of 250 μg ropeginterferon alfa-2b will be subcutaneous administrated at Day 1 visit. For patients who still have positive result (Ct <30) in SARS-CoV-2 RT-PCR at Day 15 and Day 29, the second dose of ropeginterferon alfa-2b at 350 μg and the third dose at 500 μg will be administered, respectively. For control group, patients will receive the SOC alone. The efficacy and safety of ropeginterferon alfa-2b will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 1. Willingness to provide a written ICF before entering the study;
* 2. Male or non-pregnant female patients, ≥ 18 years of age at the time of enrolment (or other age required by local regulations);
* 3. Patient with the diagnosis of COVID-19 and with the Ct value <30 in SARS-CoV-2 RT-PCR;
* 4. Patients with any comorbidity below at screening:

  1. Hematologic cancer;
  2. Solid tumor that requires chemotherapy or other systemic therapy;
  3. Well controlled autoimmune diseases; or any other medical comorbidities that requires immunosuppressive therapy;
* 5. Non-responder to the treatment of any other anti-SARS-CoV-2 drugs, i.e., remdesivir, nirmatrelvir/ritonavir, and/or molnupiravir; or patients who is not suitable to receive the other anti-SARS-CoV-2 drugs by investigator's judgement and has Ct <30 14 days after the symptom onset of COVID-19. Non-responder is defined as a patient who received remdesivir, nirmatrelvir/ritonavir, and/or molnupiravir but still has Ct <30 14 days after the symptom onset of COVID-19.
* 6. Agrees to the collection of nasopharyngeal or pharyngeal swabs and blood sample as per protocol.

Exclusion Criteria:

* 1. Known history or presence of decompensated cirrhosis of the liver (Child-Pugh B or C) before study entry;
* 2. Chronic kidney disease with eGFR <15 mL/min/1.73 m2;
* 3. Females who are breast-feeding, lactating, pregnant or intending to become pregnant;
* 4. Known history of severe allergic or hypersensitivity reactions to the active substance or to any of the excipients of ropeginterferon alfa-2b;
* 5. Known history or presence of poorly controlled or clinically significant medical conditions that are not suitable to be enrolled, at the discretion of the investigator, e.g., major psychiatric (including but not limited to those with severe depression, severe bipolar disorder, schizophrenia, suicidal ideation or history of suicidal attempt) or poorly controlled autoimmune diseases;
* 6. Clinically significant medical conditions known to interfere with absorption, distribution, metabolism or excretion of the study drugs;
* 7. Patients treated by monotherapy of telbivudine or any other combination therapy with telbivudine within 1 month prior to screening;
* 8. Use of an investigational medical product within 1 month prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2024-05-16 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Time from randomization to the achievement of Ct value ≥30 in SARS-CoV-2 quantitative reverse transcriptase polymerase chain reaction (RT-PCR) | Up to Day 57
  To compare the time from randomization to the achievement of Ct value ≥30 in SARS-CoV-2 quantitative RT-PCR between the Study and Control groups

SECONDARY OUTCOMES:
The proportion of patients who achieve Ct value ≥30 in quantitative SARS-CoV-2 RT-PCR at Day 15, Day 29, and Day 43 | Up to Day 43
  The proportion of patients who achieve Ct value ≥30 in quantitative SARS-CoV-2 RT-PCR at Day 15, 29, and 43, compared between the Study and Control groups
Change from randomization in the clinical status | Up to Day 43
  The change from randomization in the clinical status of patient on WHO clinical progression scale at Day 15, 29, and 43, compared between the Study and Control groups
Change of SpO2 | Up to Day 43
  The change of SpO2 from randomization to Day 15, 29, and 43, compared between the Study and Control groups
The occurrence and the accumulated duration (days) of supple-mental oxygen | Up to Day 57
  To compare the occurrence and the accumulated duration (days) of supplemental oxygen between the Study and Control groups
The occurrence and the accumulated duration (days) of mechanical ventilation | Up to Day 57
  To compare the occurrence and the accumulated duration (days) of mechanical ventilation between the Study and Control groups

CONTACTS AND LOCATIONS:
Overall Officials: Wang-Huei Sheng, M.D. Ph.D, Principal Investigator — Center of Infection Control of National University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu WD, Hou HA, Li KJ, Qin A, Tsai CY, Sheng WH. Study Protocol of a Randomized Controlled Clinical Trial to Evaluate the Efficacy and Safety of Ropeginterferon Alfa-2b in COVID-19 Patients with Comorbidities. Adv Ther. 2024 Feb;41(2):847-856. doi: 10.1007/s12325-023-02715-7. Epub 2023 Nov 27. PMID 38010606